CLINICAL TRIAL: NCT01695226
Title: Randomized Controlled Phase II Trial of Pre-operative Celecoxib Treatment in Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MUMC MEC 04-038
Record Dates: First submitted 2012-09-25; First posted 2012-09-27 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2012-09

CONDITIONS: Breast Neoplasms; Breast Cancer
Keywords: Celecoxib; Clinical trial, Phase II; Oligonucleotide Array Sequence Analysis
MeSH Terms: conditions — Breast Neoplasms | interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator): pre-operative placebo twice daily for two to three weeks
  Interventions: Drug: Placebo
- celecoxib (Experimental): pre-operative celecoxib (400 mg) twice daily for two to three weeks
  Interventions: Drug: celecoxib

INTERVENTIONS:
Drug: celecoxib — pre-operative celecoxib (400 mg) twice daily for two to three weeks
  Other Names: celebrex
  Arms: celecoxib
Drug: Placebo — pre-operative placebo twice daily for two to three weeks
  Arms: placebo

SUMMARY:
Cyclooxygenase-2 (COX-2) is frequently over-expressed in primary breast cancer. There is evidence that COX-2 inhibition exerts anti-tumor effects in breast cancer. To further determine the effect of COX-2 inhibition in primary breast cancer, we aimed at studying the changes in breast cancer tissues of patients treated with the selective COX-2 inhibitor celecoxib.

In a single-centre double-blinded phase II study, breast cancer patients were randomised to receive either pre-operative celecoxib (400 mg) or placebo twice daily for two to three weeks. We collected fresh-frozen pre-surgical biopsies (before treatment) and surgical excision specimens (after treatment) to assess the tumor changes by use a cDNA microarray, which allows to study the genome-wide changes at the transcriptional level.

ELIGIBILITY:
Inclusion Criteria:

* Female patients suspected of having invasive breast cancer, >1 cm in diameter, and in whom there is an indication for a core or incision biopsy
* Age <75 years at time of diagnosis
* Patient willing and able to comply with the study prescriptions
* Patient able to give written informed consent before patient registration/randomisation
* Pre- and post-menopausal patients are eligible
* Hormone receptor positive and negative patients are eligible
* A negative pregnancy test in pre-menopausal women

Exclusion Criteria:

* HIV, HBV or HCV positivity
* Known hypersensitivity to NSAIDs
* A history of upper gastro-intestinal bleeding
* Endoscopically proven upper gastro-intestinal ulceration
* Patients using NSAIDs, including salicyclic acid
* Systemic use of corticosteroids
* A history or the presence of any other malignancy excepting adequately treated squamous cell skin cancer or in situ carcinoma of the cervix
* Patients who have been treated with neo-adjuvant chemotherapy or hormone therapy

Ages: 18 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-02; Primary Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
whole-genome expression after celecoxib treatment
  Affymetrix arrays were performed on pre- and post treated (celecoxib and placebo) breast cancer tissues

SECONDARY OUTCOMES:
Percent change of Ki-67 protein positivity in celecoxib-treated breast cancer tissues versus placebo-treated tissues

OTHER OUTCOMES:
Measurement of protein expression of CD34 and CASP3 in post-treated (celecoxib and placebo) breast cancer tissues

CONTACTS AND LOCATIONS:
Overall Officials: Pierre SJ Hupperets, MD; PhD, Principal Investigator — Maastricht University Medical Centre
Locations (1):
- University Hospital Maastricht, Maastricht, Limburg, Netherlands

REFERENCES:
- [Result] Brandao RD, Veeck J, Van de Vijver KK, Lindsey P, de Vries B, van Elssen CH, Blok MJ, Keymeulen K, Ayoubi T, Smeets HJ, Tjan-Heijnen VC, Hupperets PS. A randomised controlled phase II trial of pre-operative celecoxib treatment reveals anti-tumour transcriptional response in primary breast cancer. Breast Cancer Res. 2013 Apr 8;15(2):R29. doi: 10.1186/bcr3409. PMID 23566419